CLINICAL TRIAL: NCT06404554
Title: A Prediction Model of Anastomotic Stricture After Rectal Cancer: a Retrospective Cohort Analysis
Brief Title: A Prediction Model of Anastomotic Stricture After Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Daorong Wang, Clinical Professor, Northern Jiangsu People's Hospital
Other Study IDs: NorthernJiangsu004
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer; Rectal Cancer; Anastomotic Stenosis
Keywords: nomogram; rectal cancer; anastomotic stricture
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with anastomotic stricture: without any intervention, patients diagnose as anastomotic stricture after rectal cancer surgery
  Interventions: Other: without any intervention
- patients without anastomotic stricture: without any intervention, patients does not diagnose as anastomotic stricture after rectal cancer surgery
  Interventions: Other: without any intervention

INTERVENTIONS:
Other: without any intervention — without any intervention

SUMMARY:
Background: Anastomotic stricture significantly impacts patients' quality of life and long-term prognosis. However, current clinical practice lacks accurate tools for predicting anastomotic stricture. This study aimed to develop a nomogram to predict anastomotic stricture in patients with rectal cancer who have undergone anterior resection.

Methods: 1542 eligible patients will be recruited for the study. Least absolute shrinkage selection operator (Lasso) analysis will be used to preliminarily select predictors. A prediction model will be constructed using multivariate logistic regression and presented as a nomogram. The performance of the nomogram will be evaluated using receiver operating characteristic (ROC) curves, calibration diagrams, and decision curve analysis (DCA). Internal validation will be conducted by assessing the model's performance on a validation cohort.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmation of rectal cancer;
2. eligibility for surgical intervention;
3. undergoing first rectal cancer surgery;
4. acquisition of written informed consent from patients and their families;
5. no history of hypertrophic scar or allergic predispositions.

Exclusion Criteria:

1. absence of postoperative follow-up or anastomosis details;
2. patients subjected to Hartmann or Miles procedures;
3. emergency surgery candidates due to conditions like perforation or obstruction;
4. diagnosis of multiple primary malignancies;
5. intraoperative discovery of widespread implant metastases within the abdominal cavity;
6. severe comorbidities;
7. anastomotic recurrence of rectal cancer;
8. patients who had undergone stapled hemorrhoidopexy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent anterior resection for rectal cancer at the Department of Gastrointestinal Surgery, Northern Jiangsu People's Hospital. All participants received radical treatment consistent with total mesorectal excision (TME) principles
Sampling Method: Probability Sample
Enrollment: 1542 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
patients with anastomotic stricture | up to six months
  Within six months after rectal cancer surgery, the patient was diagnosed with benign stricture of the rectal anastomosis
patients without anastomotic stricture | up to six months
  Within six months after rectal cancer surgery, the patient was not diagnosed with benign stricture of the rectal anastomosis

CONTACTS AND LOCATIONS:
Locations (1):
- Yifan Cheng, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No